CLINICAL TRIAL: NCT04121676
Title: A Phase 1 Study of AGEN2373, an Anti-CD137 Monoclonal Antibody, as Monotherapy and in Combination With AGEN1181, an Fc-Engineered Anti-CTLA-4 Monoclonal Antibody, in Patients With Advanced Cancer
Brief Title: Anti-CD137 and Anti-CTLA-4 Monoclonal Antibody in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C-1100-01
Record Dates: First submitted 2019-10-02; First posted 2019-10-10 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Advanced Cancer
Keywords: Combination Therapy; Anti-CD137; Anti-CTLA-4; Single Agent; Monotherapy; Melanoma; Cutaneous Melanoma; Solid Tumors; Advanced Cancer; Open-Label; Dose Escalation; 4-1BB
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 2-Week Monotherapy with AGEN2373 (Experimental): 3+3 Dose escalation of AGEN2373 administered by IV.
  Interventions: Drug: AGEN2373
- 3-Week Monotherapy with AGEN2373 (Experimental): 3+3 Dose escalation of AGEN2373 administered by IV.
  Interventions: Drug: AGEN2373
- 4-Week Monotherapy with AGEN2373 (Experimental): 3+3 Dose escalation of AGEN2373 administered by IV.
  Interventions: Drug: AGEN2373
- Combination Therapy with 3-week AGEN2373 Monotherapy Lead-In Combination with 6-week Botensilimab (Experimental): 3+3+3 Dose escalation of AGEN2373. AGEN2373 and botensilimab administered by IV.
  Interventions: Drug: AGEN2373; Drug: Botensilimab
- Combination Therapy with 3-week AGEN2373 in combination with 6-week Botensilimab (Experimental): 3+3+3 Dose escalation of AGEN2373. AGEN2373 and botensilimab administered by IV.
  Interventions: Drug: AGEN2373; Drug: Botensilimab

INTERVENTIONS:
Drug: AGEN2373 — An Anti-CD137 Monoclonal Antibody
  Other Names: Anti-CD137
Drug: Botensilimab — Anti-CTLA-4 Monoclonal Antibody
  Other Names: AGEN1181; Anti-CTLA-4
  Arms: Combination Therapy with 3-week AGEN2373 Monotherapy Lead-In Combination with 6-week Botensilimab; Combination Therapy with 3-week AGEN2373 in combination with 6-week Botensilimab

SUMMARY:
This study is an open-label, Phase 1, multicenter study to evaluate the safety, tolerability, PK, and PD profiles of AGEN2373 as a monotherapy and in combination with botensilimab (also known as AGEN1181), and to assess the maximum tolerated dose (MTD) in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This Phase 1 study will enroll up to approximately 200 evaluable adult patients with a histologically confirmed diagnosis of advanced cancer for which no standard therapy is available or standard therapy has failed, regardless of diagnosis and prior therapies. This also includes patients with PD-1/PD-L1 R/R melanoma. Patients may be enrolled into one of 5 treatment arms:

2-Week AGEN2373 monotherapy

3-Week AGEN2373 monotherapy

4-Week AGEN2373 monotherapy

Combination of AGEN2373 and botensilimab in patients with programmed cell death protein 1 (PD-1)/programmed death-ligand 1 (PD-L1) relapsed/refractory (R/R) melanoma.

Group 1 (Monotherapy Lead-in Combination): AGEN2373 will be administered every 3 weeks (Q3W). Starting on Cycle 4, AGEN1181 will be administered on Day 1 of every other 3-week cycle (Cycles 4, 6, 8, etc.) in combination with AGEN2373.

Group 2 (Combination): AGEN2373 will be administered Q3W in combination with botensilimab administered every other cycle.

The trial will consist of a 3+3 dose escalation that will evaluate different combination dose levels of AGEN2373 monotherapy and in combination with botensilimab. Each patient will stay on the dose level and schedule assigned at trial entry. Treatment with AGEN2373 monotherapy will be up to 2 years (i.e., maximum of 34 cycles). For combination therapy, AGEN1181 will be continued up to 1 year (i.e., maximum of 8 doses) and for AGEN2373 up to 2 years (i.e., maximum of 34 cycles), or until unacceptable toxicity, disease progression, consent is withdrawn, or any criterion for stopping the study drug or withdrawal of trial occurs.

Patients who do not complete the DLT observation period (28 days for the 2-Week and 4-Week AGEN2373 Monotherapy arms and 21 days for the 3-Week AGEN2373 Monotherapy and Combination arms) after the first dose for reasons other than DLT will be replaced.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily agree to participate by giving signed, dated, and written informed consent prior to any study specific procedures. Participation in pharmacogenomics testing is optional.
2. ≥ 18 years of age.
3. Histologically or cytologically confirmed diagnosis of a solid tumor that is currently metastatic or locally advanced for which no standard therapy is available or standard therapy has failed.
4. Measurable disease on imaging based on RECIST 1.1.
5. Life expectancy of ≥ 3 months and ECOG performance status of 0 or 1.
6. Adequate organ and bone marrow reserve function, as indicated by the following laboratory values:

   * Adequate hematological function, defined as absolute neutrophil count ≥ 1.5 × 10^9/L, platelet count ≥ 100 × 10^9/L, and hemoglobin ≥ 8 g/dL without recent transfusion (defined as a transfusion that has occurred within 2 weeks of the hemoglobin measurement)
   * Adequate liver function, defined as total bilirubin level ≤ 1.5 × upper limit of normal (ULN), aspartate aminotransferase ≤ 2.5 × ULN, and alanine aminotransferase ≤ 2.5 × ULN, albumin ≥ 3 g/dL, and alkaline phosphatase ≤ 2.5 × ULN or ≤ 5 × ULN for patients with liver metastases
   * Adequate renal function defined as creatinine ≤ 1.5 × ULN OR measured or calculated creatinine clearance ≥ 40 mL/minute per institutional standard. Assessment methods should be recorded
   * Adequate coagulation, defined as international normalized ratio or prothrombin time ≤ 1.5 × ULN and activated partial thromboplastin time ≤ 1.5 × ULN (unless patient is receiving anticoagulant therapy)
7. Patients with a history of prior malignancy are eligible if treatment was completed ≥ 2 years prior to the first dose of study treatment and the patient has no evidence of disease.
8. Patients must provide a sufficient and adequate formalin-fixed paraffin-embedded tumor tissue sample (biopsy) collected after the last dose of prior anti-cancer therapy and before the first dose of study treatment from a site not previously irradiated and agree to mandatory on-treatment biopsy if clinically feasible.
9. Female patients of childbearing potential must have a negative serum pregnancy test at screening (within 72 hours of first dose of study medication). Non-childbearing potential is defined as 1 of the following:

   * ≥ 45 years of age and has not had menses for > 1 year
   * Amenorrheic for > 2 years without a hysterectomy and oophorectomy and follicle-stimulating hormone value in the postmenopausal range upon prestudy (screening) evaluation
   * Status is post-hysterectomy, -bilateral oophorectomy, or -tubal ligation
10. Female patients of childbearing potential must be willing to use highly effective contraceptive measures starting with the Screening Visit through 90 days after last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception method for the patient.
11. Male patients with a female partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the study starting with the Screening Visit through 90 days after the last dose of study treatment is received. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner. Note: Abstinence is acceptable if this is the established and preferred contraception method for the patient.

Specific Melanoma Criteria:

Note: these specific criteria below are in addition to the general criteria above and supersede the general criteria in some cases.

Inclusion:

1. Histological confirmation of cutaneous melanoma.
2. Progression on or within 24 weeks of stopping treatment with a PD-1/PD-L1 confirmed per Society for Immunotherapy of Cancer (SITC).
3. Patients with BRAF V600-positive tumor(s) should also have received prior treatment with a BRAF inhibitor (alone or in combination with a MEK inhibitor) or have declined targeted therapy.

Note: Patients with BRAF V600-positive tumors with no clinically significant tumor-related symptoms nor evidence of rapidly progressive disease are not required to be treated with a BRAF inhibitor (alone or in combination with a MEK inhibitor) based on Investigator's decision.

Exclusion Criteria:

1. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 3 weeks of first dose of current study treatment.
2. Received prior systemic cytotoxic chemotherapy, biological therapy, radiotherapy, or major surgery outside of the acceptable washout period prior to first dose of study drug. A 1-week washout is permitted for palliative radiation to non-central nervous system (CNS) disease, with Sponsor approval.

   The following washout windows are acceptable from prior treatments (i.e., patients with time periods less than the following should be excluded):
   * Cytotoxic agent ≥ 3 weeks is acceptable (i.e., < 3 weeks should be excluded)
   * Monoclonal antibodies ≥ 4 weeks is acceptable (i.e., < 4 weeks should be excluded)
   * Proteasome inhibitors or corticosteroids ≥ 2 weeks is acceptable (i.e., < 2 weeks should be excluded)
   * Small molecule/tyrosine kinase inhibitor within 14 days or less than 5 circulating half-lives of investigational drug
   * Having a previous SARS-CoV-2 vaccine > 7 days before administration. For vaccines requiring more than 1 dose, the full series should be completed prior to Cycle 1 Day 1, when feasible, and when the delay in initiation of study treatment would not put the study patients at risk
3. Patients who have received prior anti-CD137 therapy may be enrolled upon agreement with the Sponsor.
4. Persistent toxicity of NCI-CTCAE version 5.0 Grade > 1 severity that is related to prior therapy. Note: Sensory neuropathy or alopecia of Grade ≤ 2 are acceptable.
5. Expected to require any other form of systemic or localized antineoplastic therapy while on study (including maintenance therapy with another agent, radiation therapy, and/or surgical resection).
6. History of:

   * Severe (Grade ≥ 3) hypersensitivity reactions to fully human monoclonal antibodies
   * Immune-related adverse event requiring treatment with systemic steroids for > 7 days (refer to Exclusion Criterion #7 for exceptions) excluding Grade 1 or 2 rash
   * Interstitial lung disease or lung disease which may interfere with the assessment of pneumonitis
   * Uncontrolled asthma (i.e., ≥ 3 features of partly controlled asthma)
   * Pneumonitis that has required oral or IV corticosteroids
7. Receiving systemic corticosteroid therapy per Exclusion Criterion #2, or any other form of systemic immunosuppressive medication. Note: Corticosteroid use as a premedication for IV contrast allergies/reactions is allowed. Patients who are receiving daily corticosteroid replacement therapy are also an exception to this rule. Daily prednisone at doses of ≤ 10 mg or equivalent hydrocortisone dose are examples of permitted replacement therapy. Use of inhaled or topical corticosteroids is permitted.
8. CNS tumor, metastasis(es), and/or carcinomatous meningitis identified either on the baseline brain imaging obtained during the Screening Period or identified prior to consent. Note: Patients with history of brain metastases that have been treated may participate provided they show evidence of stable supra-tentorial lesions at screening (defined as 2 brain images, both of which are obtained after treatment to the brain metastases and obtained ≥ 4 weeks apart). In addition, any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have returned to baseline or resolved. Any steroids administered as part of this therapy must be completed ≥ 3 days prior to first dose of study medication.
9. Active or history of autoimmune disease that requires systemic treatment within 2 years of the start of study treatment (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Note: Patients with autoimmune conditions requiring hormone replacement therapy or topical treatment are eligible.
10. Has had an allogeneic tissue/solid organ transplant except for corneal transplantation.
11. Active infection requiring systemic treatment.
12. Active infection with HIV and CD4+ T-cell count <350/μL. Patients not on established antiretroviral therapy for at least 4 weeks and having a detectable HIV viral load. Testing is not required for eligibility.
13. Active infection with hepatitis B (surface antigen); or infection with hepatitis C, defined by a detectable viral load. Testing is required for eligibility only if patient has a known or suspected history of infection.
14. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ II), or serious uncontrolled cardiac arrhythmia requiring medication.
15. History or current evidence of any condition, therapy, any active infections, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
16. Known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study.
17. Legally incapacitated or has limited legal capacity.
18. Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicity (DLT) | First 28 days of treatment Q2W and Q4W and First 21 days Q3W
  DLT in patient in dose escalation phase
Frequency of treatment-emergent adverse events (TEAEs) | Screening to 90 days from last dose
  According to NCI-CTCAE Version 5.0, vital signs (blood pressure, heartrate, and temperature), physical examinations, 12-lead electrocardiogram, Eastern Cooperative Oncology Group (ECOG) performance status, and clinical laboratory assessments for all dose groups
Severity of treatment-emergent adverse events (TEAEs) | Screening to 90 days from last dose
  According to NCI-CTCAE Version 5.0, vital signs (blood pressure, heartrate, and temperature), physical examinations, 12-lead electrocardiogram, Eastern Cooperative Oncology Group (ECOG) performance status, and clinical laboratory assessments for all dose groups
Duration of treatment-emergent adverse events (TEAEs) | Screening to 90 days from last dose
  According to NCI-CTCAE Version 5.0, vital signs (blood pressure, heartrate, and temperature), physical examinations, 12-lead electrocardiogram, Eastern Cooperative Oncology Group (ECOG) performance status, and clinical laboratory assessments for all dose groups

SECONDARY OUTCOMES:
Maximum observed concentration at steady state (Cmax-ss) | Day 1 of dosing through 90 days from the last dose
  PK Profile of AGEN2373 and botensilimab
Minimum observed concentration at steady state (Cmin-ss) | Day 1 of dosing through 90 days from the last dose
  PK Profile of AGEN2373 and botensilimab
Area under the plasma/serum concentration-time curve within time span t1 to t2 at steady-state (AUC(t1-t2)-ss) | Day 1 of dosing through 90 days from the last dose
  PK Profile of AGEN2373 and botensilimab
Area under the plasma/serum concentration-time curve from time zero to time t (AUC(0-t)) | Day 1 of dosing through 90 days from the last dose
  PK Profile of AGEN2373 and botensilimab
Area under the plasma/serum concentration-time curve from time zero to infinity (AUC(0-∞)) | Day 1 of dosing through 90 days from the last dose
  PK Profile of AGEN2373 and botensilimab
Time to maximum observed concentration (tmax) | Day 1 of dosing through 90 days from the last dose
  PK Profile of AGEN2373 and botensilimab
Terminal disposition rate constant (λz) | Day 1 of dosing through 90 days from the last dose
  PK Profile of AGEN2373 and botensilimab
Terminal elimination half-life (t1/2) | Day 1 of dosing through 90 days from the last dose
  PK Profile of AGEN2373
Systemic clearance (CL) | Day 1 of dosing through 90 days from the last dose
  PK Profile of AGEN2373 and botensilimab
Volume of distribution (Vd) | Day 1 of dosing through 90 days from the last dose
  PK Profile of AGEN2373 and botensilimab
Immunogenicity of AGEN2373 | Pre-dose through 3 months after the last dose
  ADA Profile of AGEN2373 and botensilimab
Overall Response Rate (ORR) | Evaluated throughout the protocol up to 2 years
  per RECIST 1.1
Duration of Response (DOR) | First observation of documented disease progression (or death within 12 weeks of the last tumor assessment)
  per RECIST 1.1
Disease Control Rate (DCR) | Time Frame: 24 weeks of first dose
  including complete and partial responders and stable disease [SD] for at least 12 weeks per RECIST 1.1
Progression Free Survival (PFS) | First treatment administration to first observation of documented disease progression (or death within 12 weeks of last tumor assessment)
  median and/or rate as defined in the statistical analysis plan

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Agenus Inc.
Locations (12):
- United States (12):
  - University of Southern California Norris Comprehensive Cancer Center/ Hoag, Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Miami, Coral Gables, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Atlantic Health System, Morristown, New Jersey
  - Roswell Park Comprehensive Cancer Care, Buffalo, New York
  - Columbia University, New York, New York
  - Providence Cancer Institute, Portland, Oregon
  - UPMC, Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - NEXT Oncology, San Antonio, Texas
  - University of Washington, Seattle, Washington